CLINICAL TRIAL: NCT02068755
Title: The Use of Blood Products in Patients Undergoing Cardiac Surgery
Brief Title: Blood Products in Cardiac Surgery
Acronym: BiCS
Status: Completed | Type: Observational
Sponsor: University of Turku (Other)
Collaborators: Finnish Red Cross Blood Service (Other); Central Finland Hospital District (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); Tampere University Hospital (Other); Kuopio University Hospital (Other); Helsinki University Central Hospital (Other); Satakunta Central Hospital (Other)
Responsible Party: Principal Investigator, Dr. Pirjo Mustonen, MD, PhD, Professor, University of Turku
Other Study IDs: BiCS
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Anemia; Renal Impairment; Thrombocytopenia
Keywords: anemia; renal impairment; thrombocytopenia; anticoagulation; Coronary bypass; Aortic valve surgery; Mitral valve surgery; red blood cell; platelet; fresh frozen plasma; octaplas
MeSH Terms: conditions — Anemia; Renal Insufficiency; Thrombocytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery: Patients who have undergone cardiac surgery

SUMMARY:
Blood transfusion is a common procedure essential for the treatment of patients undergoing cardiac surgery. Inappropriate transfusions, however, not only incur needless healthcare costs, but increase unnecessary risks due to transfusion reactions and infectious and immunomodulative causes. Safe and appropriate patient care requires evaluated blood component prescription practices.

Practically all patients undergoing cardiac surgery in Finland have a blood product booking from the Finnish Red Cross Blood Service. This registry contains large volumes of transfusion-related information on all Finnish patients undergoing cardiac surgery in Finnish centers. Participating hospitals were scattered to all geographical areas in Finland and concentrated to the most populated regions.

Data on the blood product use, laboratory findings one month pre-operatively and 12 months post-operatively were available.

Finnish hospitals have been required to provide information on hospital visits for the Finnish National Research and Development Centre for Welfare and Health for healthcare planning purposes. We used in part the original data sent by hospitals to the Finnish Hospital Discharge Register (FHDR).

DETAILED DESCRIPTION:
Registry includes

* >21 000 patients who underwent coronary bypass,
* >4500 patients with aortic valve replacement,
* >4000 mitral valve operation.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery performed in Finnish University and Central hospitals
* Blood product booking for surgery

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We collected data from patients who visited underwent cardiac surgery in Finnish hospitals during the years 2002 and 2012. Participating perform all the cardiac surgery in Finland and hospitals were scattered to all geographical areas in Finland.
Sampling Method: Non-Probability Sample
Enrollment: 31000 (Actual)
Dates: Start 2002-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Red blood cell infusions | 12 months
Platelet infusion | 12 months
Fresh frozen plasma | 12 months
Octaplas | 12 months

SECONDARY OUTCOMES:
All cause mortality | 12 months
myocardial infarction | 12 months
TIA/stroke/arterial embolism | 12
re-operation due to bleeding | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Mustonen, MD, PhD, Principal Investigator — Central Finland Central Hospital; Juhani Airaksinen, Prof, Principal Investigator — Turku University Hospital and University of Turku; Fausto Biancari, MD, PhD, Principal Investigator — Oulu University Hospital; Tuomas O Kiviniemi, Md, PhD, Principal Investigator — Turku University Hospital and University of Turku